CLINICAL TRIAL: NCT07228975
Title: Pilot, Non-pharmacological Clinical Investigation to Evaluate the Efficacy and Tolerability of a Dietary Supplement Containing EndoGen™ as an Adjunct Treatment to Current Therapy, in Endometriosis Symptoms in Fertile Women With Confirmed Diagnosis
Brief Title: Pilot Study on a Dietary Supplement With EndoGen™ as Adjunct Therapy in Women With Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endok s.r.l. (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EndOK 2023-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis
Keywords: endometriosis; Pain management; NSAIDs reduction; Parsely extract; Flavonoids; Anti-inflammatory; Dietary; Apigenin; Luteolin; rosemary extract; EndoGen; EndOK Green
MeSH Terms: conditions — Endometriosis; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MetrioFen Gocce (Experimental): EndOK Green contains EndoGen (TM)-an oral dose (10 drops per administration) twice daily of parsley extract, rosemary extract, other substances with Apigenin and Luteolin in hydro-alcoholic solution
  Interventions: Dietary Supplement: MetrioFen Gocce

INTERVENTIONS:
Dietary Supplement: MetrioFen Gocce — Solution-20 drops per day (equal to about 1 ml) on an empty stomach.

SUMMARY:
Current treatments for endometriosis, such as NSAIDs and hormone therapies, are meant for long-term use but often cause side effects, including stomach, liver, heart, and kidney issues; allergies; and hormonal problems like weight gain, acne, and bone loss. Therefore, one option being studied is a food supplement based on parsley extract (Petroselinum crispum), rosemary extract (Rosmarinus Officinalis L.), and selenium, combined with mountain celery and Vitamins B6, D, and E. The study's goal is to show improvement in pain and reduced use of NSAIDs in fertile women with endometriosis.

DETAILED DESCRIPTION:
This is a small, early-stage study designed to test whether a four-month treatment with EndOK Green-a supplement made from EndoGen (TM), a mixture based on parsley extract (Petroselinum crispum), rosemary extract (Rosmarinus Officinalis L.), and selenium-can help reduce pain and lower the need for NSAIDs in women with moderate endometriosis (classified as stage 2 to 4 by the American Fertility Society). EndOK Green extract contains natural compounds like flavonoids (apigenin and luteolin), myristicin, and apiol, which may help ease symptoms through anti-inflammatory, antioxidant, and hormone-balancing effects, with fewer side effects than standard medications. This study includes a 4-week observational run-in period designed to exclude patients who show a clinically meaningful response without receiving any additional treatment.

Following this period, the investigational product will be administered for 16 consecutive weeks. Treatment responders will be defined as patients who meet either of the following criteria during the last 4 weeks of the treatment phase, specifically during the menstrual period:

A reduction of at least 20% from baseline on the VAS100 pain scale (e.g., if baseline pain is 8, a score of 6.4 is sufficient), and/or a 50% reduction from baseline in exposure (duration or dosage) of NSAIDs or other pain relievers.

ELIGIBILITY:
Inclusion Criteria for the Initial Run-In Phase

1. Written informed consent, signed and dated personally by the patient.
2. Female between the ages of 18 and 45 (including limits), with no race limitation.
3. Documented endometriosis, confirmed by laparoscopy, ultrasound, or MRI, with or without biopsy, performed up to 36 months prior to the start of this investigation and independently of it.
4. Stable health condition and stable drug treatments within the past 2 months.
5. Endometriosis with a grade 2 (mild) to grade 4 (severe) AFSr score, whether or not treated with sex hormones, contraceptives, or any other specific treatment, stable for a minimum of 2 months. Note: In a first phase of the investigation, patients in class 2 and 3 will be recruited, while in a second phase, patients in class 4 will also be recruited.
6. 10-point Visual Analogue Scale (VAS) score of pain due to endometriosis of at least 4 for at least 2 days in the 4 weeks prior to run-in.

Inclusion criteria for treatment initiation Patients will start treatment with EndOK Green if they meet all of the following criteria.

1. Negative urine pregnancy test.
2. Difference, for at least two days, of no more than 10 in the 10-point Visual Analogue Scale (VAS) (10%) between the 4 weeks prior to the screening visit and the end of the run-in phase, provided that at least one menstruation occurred in the period.
3. No change in background therapy.

Exclusion Criteria Patients will be excluded if they meet even one of the following criteria:

1. Pregnancy, breastfeeding, or intending to become pregnant during the time this investigation will be conducted.
2. Absence of cycles for at least 3 months.
3. Previous hysterectomy or oophorectomy.
4. Pelvic inflammatory disease regardless of its etiology (Chlamydia Trachomatis, Neisseria gonorrhoeae, fungi, etc.) or presence of ovarian cysts.
5. Known hypersensitivity or allergy to the active substances and/or any component of the product under investigation.
6. Patient who has taken, within 4 weeks prior to inclusion, or is currently taking, dietary supplements for the treatment of pelvic pain or other symptoms of endometriosis.
7. Participation in any clinical study that has been ongoing or concluded for less than three months.
8. Patient with one or more psychiatric disorders, such as alcoholism, substance abuse or addictive disorder, bipolar disorder, schizophrenia, or other personality disorders.
9. Patient who, in the opinion of the gynecologist, will not be able to meet the prerequisites required for this investigation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Fertile female
Enrollment: 36 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants identified as a responder | Baseline, week 8 and week 16
  Assessed using the 10-point Visual Analogue Scale (VAS) or use of NSAIDs or pain relievers. A "Treatment responder" will be defined as a reduction from baseline of at least 20% change in the 10-point Visual Analogue Scale (VAS) in the last 04 weeks during the menstrual phase or a 50% reduction from baseline in exposure (duration or dosage) to NAIDs or pain relievers.

SECONDARY OUTCOMES:
Change from baseline in Pain Intensity using Endometriosis Health Profile (EHP)-30 Questionnaire | Baseline,week 8, week 16
  To assess the intensity of pain using the Endometriosis Health Profile (EHP)-30 Questionnaire. Scale of 0 to 100, where 0 indicates the best health status and 100 indicates the worst health status.
Change from baseline in quality of life evaluated using the Endometriosis Health Profile (EHP)-30 core questionnaire | Baseline,week 8, week 16
  To assess Quality of Life using the Endometriosis Health Profile (EHP)-30 core (30 items) questionnaire. Scale of 0 to 100, where 0 indicates the best health status and 100 indicates the worst health status.
Change from baseline in quality of life measured by the Endometriosis Health Profile (EHP)-30 modular questionnaire | Baseline,Week 8 and Week 16
  To assess quality of life using the Endometriosis Health Profile (EHP)-30 modular questionnaire. Scale of 0 to 100, where 0 indicates the best health status and 100 indicates the worst health status.
Incidence of treatment-emergent effects (Safety and Tolerability) | Baseline, week 4, week 8, week 12 and week 16
  Record of adverse events
Measurement of Adherence to treatment | Baseline,Week 4, week 8, week 12, week 16
  Compliance by self-report tool questionnaire-yes or no question on if they adhered to the treatment, and if not, what was the percentage of doses not taken, and for what reason.
Changes in NSAID or other pain medication use | Baseline, Week 4, Week 8, Week 12, Week 16
  Evaluation of pain medications (dose and/or frequency), participant diary, and use of painkillers questionnaire
Overall self-assessment of efficacy and tolerability using a 5-point scale | Week 16
  Overall efficacy and tolerability are rated on a 0 to 4 scale, with 0 being little to no effectiveness and/or tolerability and 4 being excellent effectiveness and/or tolerability.
Overall physician-assessment of efficacy and tolerability using a 5-point scale | Week 16
  Overall efficacy and tolerability are rated on a 0 to 4 scale, with 0 being little to no effectiveness and/or tolerability and 4 being excellent effectiveness and/or tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Corsetti, CEO, Study Director — ENDOK S.R.L. - Via di Valle Alessandra, 53, Rome (RM) - Italy; Luciano Serra, Chief Scientific Officer, Study Director — ENDOK S.R.L. - Via di Valle Alessandra, 53, Rome (RM) - Italy
Locations (7):
- Italy (7):
  - Site#4 - Via Nicola Tridente, 35, Bari, BA
  - Site#1 - Via Europa, 67, Alzano Lombardo, BG
  - Site#3 - Via Enrico De Nicola, 171, Camaiore, LU
  - Site#6 - Capo di piazza Gianni Bartoli, 1, Trieste, TS
  - Site#5 - Via Sabbionera, 45, Latisana, UD
  - Site#2 - Borgo Sant'Agnese, 93, Portogruaro, VE
  - Site#7 - Via S.Maria del Pozzo, 106, Somma Vesuviana

IPD SHARING:
Plan to Share IPD: No